CLINICAL TRIAL: NCT05712304
Title: Impact of the Second vs. Conventional Examination of the Proximal Colon on Adenoma Miss Rate, a Prospective Randomized Tandem Trial
Brief Title: Impact of SE of the Proximal Colon on the AMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third People's Hospital of Jingdezhen City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LL202211
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Adenoma Miss Rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional examination (No Intervention): For patients in the CE group, the colonoscope was withdrawn directly from the splenic flexure to the rectum, and polyps that were found were removed
- second examination (Experimental): For patients in the SE group, the colonoscope was reinserted into the cecum, additional polyps were removed from the proximal colon during the third withdrawall(third pass), and the remainder of the colon from splenic flexure to rectum was examined in a standard manner
  Interventions: Diagnostic Test: second examination of the proximal colon

INTERVENTIONS:
Diagnostic Test: second examination of the proximal colon — For patients in the SE group, the colonoscope was reinserted into the cecum, additional polyps were removed from the proximal colon during the third withdrawall(third pass), and the remainder of the colon from splenic flexure to rectum was examined in a standard manner
  Arms: second examination

SUMMARY:
.Studies have demonstrated that the second examination of the proximal colon can significantly increase the proximal ADR.This study aimed to determine the impact of second examination of the proximal colon on AMR compared to conventional examination.Consecutive patients aged 40-75years undergoing colonoscopy for screening.Tandem withdrawal was used in the proximal colon.Patients were randomly assigned to either the second examination(SE) or the conventional examination(CE) group.The primary outcome measure was proximal AMR,defined as the number of proximal adenomas detected in the second pass（CE group）or the third pass（SE group）divided by the total number of proximal adenomas detected during the tandem colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is routinely performed for detection and removal of colorectal adenomas, thereby preventing colorectal cancer(CRC).The adenoma miss rates(AMR) still ranges between 26%-62%,and missed adenomas may contribute to the development of interval CRC.Therefore, there is currently considerable interest in improving AMR during a colonoscopy.The second examination has recently attracted increasing attention.since it only requires a relatively short procedure time and does not require any specialized equipment.Thus, we performed an randomized controlled trial (RCT) in patients undergoing colonoscopy for screening to determine the impact of second examination of the proximal colon on AMR compared to conventional examination.

This study aimed to determine the impact of second examination of the proximal colon on AMR compared to conventional examination.Consecutive patients aged 40-75years undergoing colonoscopy for screening.Patients were excluded if they failed cecal intubation, prior colorectal resection, inadequate bowel preparation quality (Boston Bowel Preparation Scale (BBPS)scores < 2 in any segment of the colon), inflammatory bowel disease or intestinal tuberculosis, familial polyposis syndrome, coagulation dysfunction, or polyp retrieval failure.

Consecutive patients aged 40-75years undergoing colonoscopy for screening.Tandem withdrawal was used in the proximal colon.The colonoscope was inserted in a standard manner. After successful insertion in the cecum, the colonoscope was slowly withdrawn to the splenic flexure and the mucosa was carefully observed, the polyps that were found were removed for histopathologic examination(first pass).Once the splenic flexure was reached, the position of splenic flexure was marked by creating a suction mark or taking a small biopsy. Subsequently, the colonoscope was advanced to the cecum again, additional polyps were removed from the proximal colon during the second withdrawal(second pass). When the colonoscope completed the two forward view examination of the proximal colon (defined as proximal to the splenic flexure), patients were randomly assigned to either the second examination(SE) or the conventional examination(CE) group. The randomization sequence was computer-generated and concealed in sequentially numbered sealed opaque envelopes, at this moment, the envelope was opened. For patients in the SE group, the colonoscope was reinserted into the cecum, additional polyps were removed from the proximal colon during the third withdrawall(third pass), and the remainder of the colon from splenic flexure to rectum was examined in a standard manner. For patients in the CE group, the colonoscope was withdrawn directly from the splenic flexure to the rectum, and polyps that were found were removed. Multiple diminutive hyperplastic polyps (≤ 5 mm) in the sigmoid colon and rectum were not subjected to removal, and only one representative polyp biopsy was analyzed. We recorded all adverse events at the time of the colonoscopy and for one week there after The cecal intubation time and withdrawal time were recorded by an assistant with a stopwatch. The time for polypectomy and biopsy were excluded from the withdrawal time. The primary outcome measure was proximal AMR,defined as the number of proximal adenomas detected in the second pass（CE group）or the third pass（SE group）divided by the total number of proximal adenomas detected during the tandem colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients aged 40-75years undergoing colonoscopy for screening

Exclusion Criteria:

failed cecal intubation, prior colorectal resection, inadequate bowel preparation quality (Boston Bowel Preparation Scale (BBPS)scores < 2 in any segment of the colon), inflammatory bowel disease or intestinal tuberculosis, familial polyposis syndrome, coagulation dysfunction, or polyp retrieval failure.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
proximal AMR | 2 years
  the number of proximal adenomas detected in the second pass（CE group）or the third pass（SE group）divided by the total number of proximal adenomas detected during the tandem colonoscopy.

SECONDARY OUTCOMES:
proximal polyp miss rate | 2 years
  the number of proximal polyps detected in the second pass（CE group）or the third pass（SE group）divided by the total number of proximal polyps detected during the tandem colonoscopy
Per-patient proximal AMR or per-patient proximal PMR | 2 years
  the number of patients in whom proximal adenomas or polyps were detected only in the second pass（CE group）or the third pass（SE group）divided by the total number of patients with at least one proximal adenoma or polyp detected during the tandem colonoscopy
The adenoma detection rate (ADR) or polyp detection rate (PDR) | 2 years
  the proportion of patients with at least one adenoma or polyp detected during the tandem colonoscopy
Adenoma per colonoscopy (APC) or polyp per colonoscopy (PPC) | 2 years
  the total number of adenomas or polyps divided by the total number of patients
proximal advanced AMR(AAMR) | 2 years
  Advanced adenoma is defined as an adenoma with a size ≥10 mm, with tubulovillous or villous histology, or with high-grade dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: li yang, Study Director — Third People's Hospital of Jingdezhen,
Locations (2):
- China (2):
  - Second People's Hospital of Jingdezhen City, Jingdezhen, Jiangxi
  - Third People's Hospital of Jingdezhen City, Jingdezhen, Jiangxi

IPD SHARING:
Plan to Share IPD: No